CLINICAL TRIAL: NCT06101212
Title: The Predictive Effect of Impulsivity and Coping Skills on Quality of Life in Patients with Bipolar Disorder
Brief Title: Predictors of Quality of Life in Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Kubra TOHUMCU (Other)
Responsible Party: Sponsor-Investigator, Kubra TOHUMCU, principal investigator, University of Gaziantep
Organization: University of Gaziantep (Other)
Other Study IDs: Gaziantep University KBRTHMC
Record Dates: First submitted 2023-10-01; First posted 2023-10-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Quality of life; Impulsivity; Coping attitudes
MeSH Terms: conditions — Bipolar Disorder; Impulsive Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: survey — After obtaining the informed consent form, a 10-15 minute questionnaire will be applied to the patients included in the study.

SUMMARY:
This study was planned to determine the predictive effects of impulsivity and coping skills on quality of life in patients with bipolar disorder. The sample of the study, which was carried out in a descriptive design, will consist of 80 patients who applied to Adıyaman Besni State Hospital Psychiatry Outpatient Clinic with a diagnosis of bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 and who were in the euthymic period according to the doctor's control. It was planned to collect the data by applying the Personal Information Form prepared by the researchers, "Brief Quality of Life in Bipolar Disorder", "Barratt Impulsivity Scale -11 Short Form" and "Coping Attitudes Evaluation Scale". The data will be evaluated with descriptive statistics, Mann-Whitney U-test, Kruskal Wallis test, Pearson correlations and regression analyses using Statistical Package for the Social Sciences 22 software. Scale use and ethics committee permission were obtained from the responsible authors of the scales before the study.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic illness characterised by periods of illness and recovery, which can cause significant psychosocial impairment and disability. It affects more than 1% of the world population regardless of demographic characteristics such as ethnicity, nationality, socioeconomic status and is one of the leading causes of global disability. Bipolar disorder can cause serious cognitive and functional impairments and maintaining life with this disorder involves some difficulties for the individual. Functional impairments such as deterioration in family relationships, problems in work life and incompatibilities in social relationships negatively affect both the well-being and quality of life of the individual. Many individuals diagnosed with bipolar disorder have functional disorders that can cause low quality of life. Quality of life is recognised as an important outcome measure for the effectiveness of treatment of mental disorders. Compared to healthy individuals, the quality of life of patients with bipolar disorder is significantly impaired in both the euthymic and symptomatic periods. The ability to cope with difficulties is assumed to be a protective factor for quality of life. However, individuals diagnosed with bipolar disorder are exposed to more stressful events due to their illness and experience coping problems, including in the euthymic period. For these reasons, developing coping skills is among the targets in the treatment process of bipolar disorder. The stress coping strategies of these individuals may even affect the risk of suicide. Bipolar disorder is a serious illness that causes increased mortality, including death by suicide. Approximately 10-20% of these individuals end their lives and approximately one third of these individuals attempt suicide at least once.

Patients with bipolar disorder and previous suicide attempts have a worse quality of life. One of the most important factors associated with suicide and morbidity in bipolar disorder is impulsivity. Impulsivity, which can be defined as a predisposition to unplanned reactions to internal and external stimuli regardless of negative consequences and the absence of behavioural inhibition, is one of the clinical features of bipolar disorder. Although it is more common during manic episode, it can also be found in other mood phases. Bipolar disorder is characterised by high impulsivity even during recovery periods. Increased impulsivity is not only associated with suicide attempts but may also lead to functional impairment. Impulsive behaviours may cause long-term negative consequences in bipolar disorder that may affect quality of life. In the literature, it has been revealed that high impulsivity is associated with poor quality of life.

In the light of this information, this study aimed to determine the predictive effects of impulsivity and coping skills on quality of life in patients with bipolar disorder.

METHOD Sample The descriptive study is planned to be conducted in Adıyaman Besni State Hospital between October 2023-February 2024. The population of the study will consist of individuals who applied to the Psychiatry Outpatient Clinic of Adıyaman Besni State Hospital on the dates of the study, who received outpatient treatment with the diagnosis of bipolar according to Diagnostic and Statistical Manual of Mental Disorders-5 and who were in the euthymic period according to the doctor's control. G* Power programme was used to calculate the sample size. The confidence interval α=0.05, the power of the test (1-β) 0.95, the effect size dz= 0.5 were calculated as a total of 54 people (presented in the appendix).

The data will be collected by researcher Kubra Tohumcu through face-to-face interview technique. The patients constituting the sample of the study will be directed to the researcher by the outpatient clinic doctor. The data were planned to be collected by applying the "Personal Information Form", "Brief Quality of Life in Bipolar Disorder Scale", "Barratt Impulsivity Scale -11 Short Form" and "Coping Attitudes Evaluation Scale" prepared by the researchers.

Individual Information Form: This form, organised by the researchers, included 17 questions to determine the demographic information of the participants.

Brief Quality of Life in Bipolar Disorder Scale: Developed in 2010 by Michalak and Murray, the Turkish validity and reliability study of the scale was conducted by Gümüş et al. It is a 5-point Likert-type scale (1=Strongly Disagree, 5=Strongly Agree) consisting of a total of 7 items. The total score range that can be obtained from the scale varies between 12-60. Higher scores obtained from the scale indicate a better quality of life. Cronbach Alpha internal consistency coefficient was reported as .86.

Barratt Impulsivity Scale -11 Short Form: The scale consists of a total of 15 items and three subscales. These subscales are lack of planning, motor impulsivity and attention impulsivity. The items in the scale are evaluated using a 4-point Likert-type scale (1=rarely/never, 4=almost always/always). The high scores obtained from the scale indicate a high level of impulsivity. The Cronbach's alpha internal consistency coefficient for the entire scale adapted into Turkish was reported as .82, .80 for the failure to plan subscale, .70 for the motor impulsivity subscale, and .64 for attention impulsivity.

Coping Attitudes Rating Scale: The scale is a 4-point Likert-type scale (1=I Never Do This, 4=I Mostly Do This) consisting of 5 factors and 32 items. The score range to be obtained from the scale varies between 32-128, and the high score obtained from the scale indicates that the coping attitude level is high, while the low score obtained indicates that the coping attitude level is low. In the Turkish validity and reliability study of the scale, cronbach alpha value was .766.

Data analysis: The data of the study will be evaluated using descriptive statistical methods (frequency, mean), t-test, one way Analysis of Variance, correlation and regression analyses in Statistical Package for the Social Sciences 22 package programme.

ELIGIBILITY:
Inclusion Criteria:

* Receiving outpatient treatment with a diagnosis of Bipolar Disorder according to DSM-5
* Being in euthymic mood according to the doctor's control at the time of the interview
* Having no problem in understanding and speaking Turkish
* Being in the 18-65 age group

Exclusion Criteria:

* Presence of serious sensory and cognitive impairment that would prevent answering the questionnaire
* Refusing to participate in the study after being informed
* Having another psychiatric diagnosis in addition to the diagnosis of bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The descriptive study is planned to be conducted in Adıyaman Besni State Hospital between October 2023-February 2024. The population of the study will consist of individuals who applied to the Psychiatry Outpatient Clinic of Adıyaman Besni State Hospital on the dates of the study, who received outpatient treatment with the diagnosis of bipolar according to Diagnostic and Statistical Manual of Mental Disorders-5 and who were in the euthymic period according to the doctor's control. G* Power programme was used to calculate the sample size. The confidence interval α=0.05, the power of the test (1-β) 0.95, the effect size dz= 0.5 were calculated as a total of 54 people (presented in the appendix).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
The Predictive Effect of Impulsivity on Quality of Life in Patients with Bipolar Disorder | 15 October 2023-1 February 2024
  The effect of impulsivity level on quality of life in bipolar disorder patients.
  It was planned to collect the data by applying the "Personal Information Form", "Quality of Life in Bipolar Disorder Scale Short Form", "Barratt Impulsivity Scale -11 Short Form" and "Coping Attitudes Assessment Scale" prepared by the researchers. Barratt Impulsivity Scale minimum score=15 and maximum score=60. High scores indicate high impulsivity level of individuals. The results will be evaluated in line with the data obtained.

SECONDARY OUTCOMES:
The Predictive Effect of Coping Skills on Quality of Life in Patients with Bipolar Disorder | 15 October 2023-1 February 2024
  The effect of coping skill level on quality of life in patients with bipolar disorder.
  It was planned to collect the data by applying the "Personal Information Form", "Quality of Life in Bipolar Disorder Scale Short Form", "Barratt Impulsivity Scale -11 Short Form" and "Coping Attitudes Assessment Scale" prepared by the researchers. The minimum score of the Coping Attitudes Assessment Scale=32 and the maximum score=128. High scores indicate that the coping attitude level of individuals is increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Besni State Hospital, Besni, Adıyaman Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No